CLINICAL TRIAL: NCT04859101
Title: Post-operative Sore Throat and Gum Chewing for Long Duration LMA Use: A Randomized Controlled Trial
Brief Title: Post-operative Sore Throat and Gum Chewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ANES-2021-29683
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia; Surgery
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gum (Experimental): Group 1 will receive gum immediately prior to transport to the operating room. They will be asked to chew the gum for 2 minutes and then spit the gum in the garbage.
  Interventions: Other: Gum
- Control (Other): Group 2 will not receive any gum. They will be asked to swallow twice and have no other intervention.
  Interventions: Other: Control

INTERVENTIONS:
Other: Gum — 2 minutes of gum chewing prior to procedure
  Arms: Gum
Other: Control — 2 swallows prior to procedure
  Arms: Control

SUMMARY:
The purpose of this study is to determine if chewing gum immediately prior to transport to the operating room reduces the severity of post-operative sore throat in patients who have an LMA (laryngeal mask airway) placed for procedures with duration greater than 1 hour.

DETAILED DESCRIPTION:
Patients will be randomized into two groups. Group 1 will receive a piece of gum immediately prior to transport to the operating room. They will be asked to chew the gum for 2 minutes and then spit the gum in the garbage. Group 2 will not receive any gum. They will be asked to swallow twice and have no other intervention.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient ambulatory surgery
* General anesthesia utilizing a laryngeal mask airway
* Greater than 1 hour duration

Exclusion Criteria:

* Chronic laryngitis
* Chronic bronchitis
* Asthma
* Gastroesophageal reflux disease
* Smoking within the last week
* Non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe Post-operative Sore Throat within 24 hours | 24 hour
  Moderate to severe post-operative sore throat defined as greater than 3 on an 11-point Numeric Rating Scale; 0 being no sore throat, 10 being maximum imaginable sore throat

SECONDARY OUTCOMES:
Satisfaction with Anesthesia | 24 hour
  5-point likert scale; very satisfied, satisfied, neutral, dissatisfied, very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Jacob L Hutchins, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No